CLINICAL TRIAL: NCT02984228
Title: The Efficacy of Ultrasound Guided Glenohumeral Joint Injections of Platelet Rich Plasma (PRP) Versus Hyaluronic Acid (HA) in the Treatment of Glenohumeral Osteoarthritis: a Randomized, Double-blind Control Trial
Brief Title: Platelet-rich Plasma vs. Hyaluronic Acid for Glenohumeral Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-188
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis; Shoulder Pain
MeSH Terms: conditions — Osteoarthritis; Shoulder Pain | interventions — Hyaluronic Acid; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Platelet-rich plasma (PRP) (Active Comparator): Patients will receive an injection of PRP.
  Interventions: Biological: PRP; Device: Ultrasound
- Hyaluronic Acid (Active Comparator): Patients will receive an injection of hyaluronic acid.
  Interventions: Drug: Hyaluronic Acid; Device: Ultrasound

INTERVENTIONS:
Biological: PRP
  Arms: Platelet-rich plasma (PRP)
Drug: Hyaluronic Acid
  Arms: Hyaluronic Acid
Device: Ultrasound

SUMMARY:
This study seeks to expand the current literature in demonstrating potentially efficacious, conservative treatments in the management of glenohumeral osteoarthritis (OA) and will compare ultrasound-guided injections of hyaluronic acid vs. platelet-rich plasma. We aim to obtain information measuring potential benefits of these interventions and to observe for any adverse events.

DETAILED DESCRIPTION:
Glenohumeral OA accounts for approximately 2-5% of all chronic shoulder pain and may be classified into primary and secondary forms. Primary glenohumeral OA is caused by degenerative joint disease, inflammatory arthropathies, and neuropathic arthropathy secondary to syringomyelia or diabetes. Secondary glenohumeral OA is caused by trauma, postoperative changes after arthroscopy or capulorraphy, and osteonecrosis. Hyaluronic acid is found in synovial joint fluid and has viscoelastic, chondroprotective, and possibly anti-inflammatory properties. It has been shown to increase joint lubrication. Platelet-rich plasma contains growth factors that have been shown to promote tissue regeneration. The aim of this study is to determine whether injections of hyaluronic acid or platelet-rich plasma can be used reliably to decrease pain, restore function, and improve quality of life in patients suffering from glenohumeral OA. Patients will be randomized to receive either an injection of hyaluronic acid or an injection of platelet-rich plasma. Outcomes will be assessed via questionnaires for up to 52 weeks post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* English speaking/literate
* Age 18-100 years
* Visual analog score pain >= 5
* Greater than or equal to 3 months of pain after onset of symptoms that has failed conservative treatments
* Confirmation of glenohumeral OA via routine imaging (MRI and x-ray; must be recent and within the past year)
* Transient relief of symptoms after diagnostic intra-articular injection into the glenohumeral joint

Exclusion Criteria:

* Non-English speaking/illiterate
* Painful active, concurrent cervical spine conditions
* Current non-steroidal anti-inflammatory drug (NSAID) use
* History of taking coumadin or similar anticoagulant, have a known coagulopathy, bleeding dyscrasia, or platelet count < 150,000/cubic mm
* Allergic reaction to poultry or previous viscosupplementation
* Involved in workers' compensation or active litigation involving affected shoulder
* Inability to refrain from NSAID use for 5 days prior to and 6 weeks after injection
* History of corticosteroid injection to affected shoulder within the last 3 months
* History of viscosupplementation or platelet-rich plasma to affected shoulder within the last 6 months
* Presence of acute fracture
* History of shoulder tumor
* Known uncontrolled systemic illness (uncontrolled diabetes, human immunodeficiency virus, vasculitis, autoimmune/inflammatory disease)
* Psychiatric and somatoform disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kirschner, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet-rich Plasma (PRP): Patients will receive an injection of PRP.
  PRP
  Ultrasound
- Hyaluronic Acid: Patients will receive an injection of hyaluronic acid.
  Hyaluronic Acid
  Ultrasound
Period: Overall Study
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
Started | 34 | 36
Completed | 34 | 35
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (11.5) | 68.4 (11.9) | 68.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 33 | 35 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70
Severe osteoarthritis [Count of Participants; unit: Participants] — Severity of osteoarthritis was determined from radiographs, magnetic resonance imaging, or computed tomography scans by a fellowship-trained musculoskeletal radiologist. Severe osteoarthritis was defined as severe joint space loss with formation of osteophytes (bone spurs).
  Participants | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Pain and Disability Index (SPADI) Score
Description: Score ranges from 0-100, with a higher score representing higher disability.
Time Frame: Up to 52 weeks post-procedure
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
Number analyzed (Participants) | 34 | 35
score on a scale | 50.3 [38.7 to 62] | 49 [38 to 60.5]

2. Secondary Outcome: Shoulder Function
Description: Shoulder function will be assessed using the American Shoulder and Elbow Surgeons Society Standardized Shoulder Assessment (ASES) Form. The ASES forms includes questions about difficulty performing different functions, such as putting on a coat and sleeping on the affected side. Scores range from 0 to 100, with a higher score indicating higher function and a lower score indicating lower function.
Time Frame: Up to 52 weeks post-procedure
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
Number analyzed (Participants) | 34 | 35
score on a scale | 57.8 [47.9 to 68] | 59 [46.3 to 68.5]

3. Secondary Outcome: Number of Patients Who Were Satisfied After Treatment
Description: Satisfaction will be assessed using the North American Spine Society Patient Satisfaction Index. Patients were asked to select one of the following in regards to the procedure: "The procedure met my expectations"; "The procedure improved my condition enough so that I would go through it again for the same outcome"; "The procedure helped me, but I would not go through it again for the same outcome"; or "I am the same or worse compared to before the procedure". Responses of "The procedure met my expectations" and "The procedure improved my condition enough so that I would go through it again for the same outcome" were considered to be "satisfied". The other two responses were considered to be "not satisfied".
Time Frame: Up to 52 weeks post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
Number analyzed (Participants) | 34 | 35
Participants | 20 | 20

4. Secondary Outcome: Number of Patients With Complication Events After the Procedure
Description: Any complications reported were collected. Complications include bleeding from the injection site, prolonged swelling, infection, weakness of the muscles surrounding the injected joint, and allergic reactions. Total number of available events was calculated by multiplying the number of patients with the number of follow-up time points. The percentage of complication events was calculated by summing the number of complication events and dividing that by the total number of available events, and then multiplying by 100.
Time Frame: Up to 52 weeks post-procedure
Measure: Number; unit: participants
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
Number analyzed (Participants) | 34 | 35
participants | 11 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year.
Description: Adverse events included bleeding from the injection site, swelling, infection, allergic reactions, weakness of the muscle surrounding the infected joint. The adverse event percentages noted in this section do not match the ones reported under Outcome Measures, as the Outcome Measures represent the percentage of adverse event cases among all events available (e.g., number of patients * number of follow-up time points).
Arm/Group | Platelet-rich Plasma (PRP) | Hyaluronic Acid
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 11/34 | 13/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Platelet-rich Plasma (PRP) (N=34) | Hyaluronic Acid (N=35)
Weakness of muscle surrounding injection site (Musculoskeletal and connective tissue disorders) | 9 | 9
Allergic reaction with itchiness (Immune system disorders) | 1 | 4
Infection (Infections and infestations) | 0 | 2
Difficulty moving affected shoulder joint (Musculoskeletal and connective tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02984228/Prot_SAP_000.pdf